CLINICAL TRIAL: NCT01784601
Title: Incidence of Hemidiaphragmatic Palsy After Single Shot Interscalene Block for Pain Relief in Shoulder Surgery
Brief Title: Incidence of Hemidiaphragmatic Palsy After Interscalene Block
Status: Suspended | Type: Observational
Why Stopped: Lack of human resources
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shalini Dhir, Associate Professor, Department of Anaesthesia, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 103337
Record Dates: First submitted 2013-02-01; First posted 2013-02-06 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Phrenic Nerve Paralysis
Keywords: Interscalene block; Hemidiaphragm palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control Group: We will be including all patients undergoing shoulder surgery not scheduled for a nerve block.
- Study Group: We will be including all patients undergoing shoulder surgery scheduled for a nerve block.

SUMMARY:
Primary objective of this study is to find out the incidence of hemi-diaphragmatic palsy associated with interscalene block done under ultrasound guidance.

Primary hypothesis:

• There is an incidence of hemidiaphragmatic palsy ranging fron 33-100 % after an interscalene block.

Secondary hypothesis

* The incidence of hemidiaphragmatic palsy is much less than 33% when the block is done using ultrasound.
* The incidence of hemi-diaphragmatic palsy is directly proportional to volume of local anaesthetic injected.
* The incidence of hemi-diaphragmatic palsy is directly proportional to concentration of local anaesthetic injected.

DETAILED DESCRIPTION:
Patients of either sex belonging to American Society of Anesthesiologists status 1-3 scheduled for elective shoulder surgery as an outpatient basis, planned for an interscalene block will be included in this study over a period of one year.

Potential patients will be identified from the surgeons' list. The PI or one of the co-investigators will contact them in the surgical day care in the morning of surgery and will be given information about the study. Documented informed consent will be obtained.

After obtaining informed consent, they will be examined for their diaphragm position using an ultrasound prior to block placement .

All patients will have the block initiated in the block room using standard monitors and sedation as per the standard practice in this hospital.

The patients will undergo an ultrasound examination for their diaphragm position 5 mins and 10 mins after the completion of the nerve block. Ipsilateral ( same side as the block) and contralateral ( opposite side of block) hemi-diaphragmatic excursion will be measured with the patients in supine position during quiet inspiration ,deep inspiration and forceful sniff.

In addition, bedside spirometry using a compact spirometer will be performed and FVC, FEV1 and PEFR measurements will be performed.The oxygen saturation and any evidence of dyspnea or shortness of breadth will be noted at the above mentioned intervals after the completion of the block.

All patients will receive general anesthesia in the operating room. The patient will receive IV opioids during the procedure if required.

The above mentioned data will be collected postoperatively in the recovery room 30 mins, after arrival.

ELIGIBILITY:
Inclusion Criteria:

Control Group:

Age between 18 - 80 years old Elective shoulder surgery Same day discharge Inform consent signed

Exclusion Criteria:

Ongoing Major psychiatric problems Narcotic Abuse/ Drug dependency Mental impairment / inability to cooperate with postoperative evaluation/Inability to give informed consent

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Control Group:
  We will be including all patients undergoing shoulder surgery not scheduled for a nerve block.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary outcome of this study is to find out the incidence of hemi-diaphragmatic palsy associated with interscalene block done under ultrasound guidance. Primary hypothesis: | 1 year
  We intend to scan all patients undergoing ISB who consent to be part of the study, for the diaphragm excursion to find out the incidence at our institute.

SECONDARY OUTCOMES:
In addition we will also do Spirometric analysis and assess for symptomatic respiratory insufficiency/ distress. Thus we can find the incidence of clinically significant hemi-diaphragmatic palsy. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Dhir, FRCPC, Principal Investigator — St. Joseph's Health Care
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada